CLINICAL TRIAL: NCT05423366
Title: Comparative Effects of Large Focused and Controlled Unfocused (Radial) Extracorporeal Shock Wave Therapies in the Treatment of Patellar Tendinopathy.
Brief Title: Comparative Effects of Focused and Unfocused (Radial) ESWT in the Treatment of Patellar Tendinopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Van YüzüncüYıl
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Patellar Tendinitis
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Large-Focused Extracorporeal Shock Wave Therapy (Active Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)
- Controlled-Unfocused (Radial) Extracorporeal Shock Wave Therapy (Active Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)
- Sham Extracorporeal Shock Wave Therapy (Sham Comparator)
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy (ESWT) — The ESWT device is product of Elettronica Pagani, Italy.

SUMMARY:
There is no scientific study in the literature regarding the use of different extracorporeal shock wave therapies (ESWT) in the treatment of patellar tendinopathy. In this study, we aim to investigate both the effectiveness of ESWT and which type of ESWT can be more effective in the treatment of patellar tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Engaging in active sports, being 18 years or older, history of activity-related knee pain in the patellar tendon or patellar insertion, symptoms lasting longer than 8 weeks (non-acute), VISA-P score less than 80 before treatment, pain during knee loading on tendon or tendon it remains isolated in the limited part of the bone junction and does not spread to the entire patellar region (to differentiate patellar tendinopathy and patellofemoral pain).

Exclusion Criteria:

* Being under the age of 18, acute knee or acute patellar tendon injury, chronic inflammatory joint diseases (rheumatoid arthritis, etc.), using immunosuppressive or corticosteroid medication in the last 6 months, previous knee surgery (in the anterior cruciate ligament or patellar tendon), knee in the last 1 month local (corticosteroid) injection, contraindications for ESWT treatment (eg pregnancy, malignancy, coagulopathy), previous ESWT treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | at baseline.
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse
Visual Analogue Scale (VAS) | 3 weeks after baseline.
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse
Visual Analogue Scale (VAS) | 7 weeks after baseline.
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse
Visual Analogue Scale (VAS) | 15 weeks after baseline.
  patient's self-assessment of pain, in the range of 0 to 10, higher scores mean a worse
Victorian Institute of Sports Assessment-Patella (VISA-P) | at baseline.
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. Theoretically, a maximum score of 100 and a minimum score of 0 can be obtained in the VISA-P questionnaire. Scores below 80 are usually indicative of patellar tendinopathy.
Victorian Institute of Sports Assessment-Patella (VISA-P) | 3 weeks after baseline.
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. Theoretically, a maximum score of 100 and a minimum score of 0 can be obtained in the VISA-P questionnaire. Scores below 80 are usually indicative of patellar tendinopathy.
Victorian Institute of Sports Assessment-Patella (VISA-P) | 7 weeks after baseline.
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. Theoretically, a maximum score of 100 and a minimum score of 0 can be obtained in the VISA-P questionnaire. Scores below 80 are usually indicative of patellar tendinopathy.
Victorian Institute of Sports Assessment-Patella (VISA-P) | 15 weeks after baseline.
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. Theoretically, a maximum score of 100 and a minimum score of 0 can be obtained in the VISA-P questionnaire. Scores below 80 are usually indicative of patellar tendinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Şah, Principal Investigator — Yüzüncü Yıl Üniversitesi Tıp Fakültesi
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No